CLINICAL TRIAL: NCT01006044
Title: Prospective, Phase II Clinical Trial to Evaluate Efficacy and Safety of Autologous Dendritic Cell Vaccination in Glioblastoma Multiforme Patients After Complete Surgical Resection With Fluorescence Microscope
Brief Title: Efficacy & Safety of Autologous Dendritic Cell Vaccination in Glioblastoma Multiforme After Complete Surgical Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEND/GM; 2009-009879-35 (EudraCT Number)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma multiforme, vaccine, dendritic cells, glioma
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccination (Experimental): Autologous Dendritic cells loaded with tumor lysate
  Interventions: Biological: autologous dendritic cells

INTERVENTIONS:
Biological: autologous dendritic cells — Patients will receive standard first-line therapy (surgery before radio-chemotherapy) along with the experimental treatment. The experimental treatment consists in subcutaneous vaccination with a suspension of autologous dendritic cells (cells from the same patient) produced by cell culture from monocytes from the same patient extracted by leukapheresis and pulsed with a lysate of the patient´s tumoral tissue. The first four vaccines will be administered on a monthly basis, concomitantly with the standard chemo and radiotherapy treatments, the next four vaccines, every other month and the four last vaccinations every three months.The results obtained will be compared with those of an historical control study, where patients received a standard treatment without the experimental vaccine.

SUMMARY:
1. Primary outcome measure:

   a.Evaluation of the treatment impact on progression-free survival.
2. Secondary outcome measures:

   1. Safety evaluation.

      * Direct effects attributable cell obtaining and administration.
      * Adverse events during treatment.
      * Neurological deterioration quantified using the NIH Stroke Scale.
      * Autoimmune phenomena.
   2. Evaluation of impact on other efficiency clinical parameters.

      * Overall survival.
      * Quality of life measured with EORTC questionnaire.
   3. Study of specific immune response and correlates with clinical outcome.

      * Delayed hypersensitivity.
      * Humoral response to autologous tumor cells/tumoral lysate.
      * Cellular response (proliferation, cytokine production, specific cytotoxicity).
   4. Cell line characterization and correlate the final product with clinical efficacy.

      * Phenotypic studies.

DETAILED DESCRIPTION:
A prospective, open-label, unicentric phase II trial, historical control and non-randomized.

The study will try to evaluate the efficiency and safety of the experimental treatment using a cell therapy product (tumor lysate-pulsed autologous dendritic cell vaccine) in patients with glioblastoma multiforme in whom a gross total resection is feasible. Patients will receive standard first-line therapy (surgery before radio-chemotherapy) along with the experimental treatment. The experimental treatment consists in subcutaneous vaccination with a suspension of autologous dendritic cells (cells from the same patient) produced by cell culture from monocytes from the same patient extracted by leukapheresis and pulsed with a lysate of the patient´s tumoral tissue. The first four vaccines will be administered on a monthly basis, concomitantly with the standard chemo and radiotherapy treatments, the next four vaccines, every other month and the four last vaccinations every three months.The results obtained will be compared with those of an historical control study, where patients received a standard treatment without the experimental vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of glioblastoma that have not received any previous chemotherapy or radiotherapy treatment.
* Patients are able to give informed consent and willing to comply with the protocol requirements during the study period.
* Age between 18 and 70 years
* Negative pregnancy test In female fertile subjects
* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Complete/Total resection of tumour with surgery guided by fluorescence microscopy and 5-aminolevulinic acid, observed with post operative magnetic resonance imaging. The residual lesion must be null or ≤ 1 cm3 by contrast capturing.
* Enough tumor tissue available for the cellular vaccine elaboration

Exclusion Criteria:

* Patients with infections, severe diseases or hepatic, renal or medullary failures, that in the investigator's opinion, are not eligible to participate in the study.
* Participation in other clinical trial. If the patient has participated in other clinical trial within previous months, the patient has to complete the washout period required by de the investigator.
* Patients with diagnosis of other neoplasia, except basal cell or squamous cell skin, carcinoma in situ of the cervix properly treated or other tumour curatively treated and no evidence of relapse for at least 3 years. Those cases with coexisting tumours of long-term survival prediction will be considered individually.
* Pregnant or breast-feeding women.
* Patients who need immunosuppressive drugs.
* Positive serology for HIV , hepatitis B (HBsAg) or hepatitis C virus.
* Impossible to get enough material for at least 6 cellular vaccine production.
* Absolute contraindication for the patient to receive other steps of standard treatment of glioblastoma (surgery, radio and chemotherapy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the treatment impact on progression-free survival | 5 years

SECONDARY OUTCOMES:
Safety evaluation | 5 years
  1. Direct effects attributable cell obtaining and administration
  2. Adverse events during treatment
  3. Neurological deterioration quantified using the NIH Stroke Scale
  4. Autoimmune phenomena
Evaluation of impact on other efficiency clinical parameters | 5 years
  1. Overall survival
  2. Quality of life measured with EORTC questionnaire
Study of specific immune response and correlates with clinical outcome | 5 years
  1. Delayed hypersensitivity
  2. Humoral response to autologous tumor cells/tumoral lysate
  3. Cellular response (proliferation, cytokine production, specific cytotoxicity)
Cell line characterization and correlate the final product with clinical efficacy | 5 years
  a. Phenotypic studies

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Prosper, MD, PhD, Study Director — Clinica Universidad de Navarra
Locations (1):
- Clínica Universidad de Navarra, Pamplona, Pamplona, Spain

REFERENCES:
- [Background] Liau LM, Black KL, Prins RM, Sykes SN, DiPatre PL, Cloughesy TF, Becker DP, Bronstein JM. Treatment of intracranial gliomas with bone marrow-derived dendritic cells pulsed with tumor antigens. J Neurosurg. 1999 Jun;90(6):1115-24. doi: 10.3171/jns.1999.90.6.1115. PMID 10350260
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Omuro AM, Faivre S, Raymond E. Lessons learned in the development of targeted therapy for malignant gliomas. Mol Cancer Ther. 2007 Jul;6(7):1909-19. doi: 10.1158/1535-7163.MCT-07-0047. PMID 17620423
- [Derived] Inoges S, Tejada S, de Cerio AL, Gallego Perez-Larraya J, Espinos J, Idoate MA, Dominguez PD, de Eulate RG, Aristu J, Bendandi M, Pastor F, Alonso M, Andreu E, Cardoso FP, Valle RD. A phase II trial of autologous dendritic cell vaccination and radiochemotherapy following fluorescence-guided surgery in newly diagnosed glioblastoma patients. J Transl Med. 2017 May 12;15(1):104. doi: 10.1186/s12967-017-1202-z. PMID 28499389